CLINICAL TRIAL: NCT01363141
Title: Effects of Glycooxidative Stress on Human Aging- Study #3
Brief Title: Effect of a Low Advanced Glycation End Products (AGE) Diet in the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 03-0116-3; 2R01DK091231-07A2 (NIH)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome
Keywords: Cardiovascular Diseases; Type 2 Diabetes Mellitus; Abdominal Fat; Atherogenic Dyslipidemia; Hypertension; Hyperglycemia; Insulin Resistance; Thrombosis state
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypertension; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular AGE Diet (Active Comparator): Regular AGE Diet
  Interventions: Other: Regular AGE Diet
- Low AGE Diet (Active Comparator): One year reduction in dietary AGE intake
  Interventions: Other: Low AGE Diet

INTERVENTIONS:
Other: Regular AGE Diet — Regular AGE Diet
  Arms: Regular AGE Diet
Other: Low AGE Diet — One year reduction in dietary AGE intake.
  Arms: Low AGE Diet

SUMMARY:
The investigators have previously demonstrated that Advanced Glycation End products (AGEs) are associated with several chronic diseases in humans and that blood AGE levels can be significantly reduced by simply changing the way food is cooked.

This is an interventional-randomized study in which we are trying to determine whether a diet low in AGE followed for 1 year can effectively reduce circulating AGE levels as well as markers of the metabolic syndrome in a group of patients with these abnormal markers.

DETAILED DESCRIPTION:
The metabolic syndrome (MetSyn), a well-defined cluster of pathogenic conditions, includes glucose intolerance, insulin resistance (pre-diabetes), hypertension, abdominal obesity, and dyslipidemia. The MetSyn has a strong inflammatory component and raises the risk for cardiovascular disease (CVD) by five-fold and of diabetes by two fold in aging. Although, excessive caloric intake, i.e. "over nutrition" is known to be involved in developing the MetSyn, the actual causative agents of MetSyn in human nutrition have not been determined.

The investigators have previously shown that Advanced Glycation End products (AGEs) can induce oxidant stress and inflammatory responses and modulate insulin signaling in animal models and more recently in humans. These studies separated the effects of "over-nutrition" from the pro-inflammatory effects of AGEs, a factor not previously considered. These data support our hypothesis that AGE-restriction could be an important intervention in the MetSyn in aging.

The investigators would like to demonstrate that this safe, practical and economical intervention can arrest the progression of three major "epidemics" of aging: diabetes, obesity, and vascular disease associated with the metabolic syndrome. This simple intervention could have significant health and economic implications.

Our hypothesis is that dietary AGE restriction can reverse several cardinal manifestation of the MetSyn, specifically insulin resistance, abdominal obesity and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking adult subjects with at least three of the following five characteristics of the metabolic syndrome (MetSyn):

  * Waist circumference:

Men: > 102 cm Women: > 88 cm

* Blood pressure: > 130/85 mm Hg (or use of anti-Blood Pressure medication)
* HDL-cholesterol:

Men: < 40 mg/dL Women: < 50 mg/dL

* Triglycerides: > 150 mg/dL (or use of medications for high triglycerides such as fibrates or nicotinic acid)
* Fasting blood sugar > 100 mg/dl (or use of metformin), but a Glycated hemoglobin (HbA1c) <6.5%

  * Any gender and race 50 years old or above
  * Dietary AGE intake > 12 AGE Eq/day

(Before randomization all participants will be screened with a 3-day food record and 7-day food frequency questionnaire (AGE Quick Score) to determine their average spontaneous daily intake of AGEs. Only those subjects whose daily intake is > 12 AGE Eq/day will participate in the study.)

Exclusion Criteria:

* Diagnosis of diabetes (HbA1C > 6.5 %)
* Glomerular Filtration Rate (GFR) less than 60 ml/min
* Any major cardiovascular event within the preceding 3 months
* Inability to understand or unwillingness to follow study diets
* Any unstable medical condition requiring medication adjustment or treatment within the preceding 3 months
* Any severe illness with an expected participant survival less than 1 year
* Diagnosis of HIV
* Currently receiving treatment for any inflammatory condition
* Currently receiving cancer treatment, such as radiation, chemotherapy, hormone therapy, or stem cell transplant
* Currently participating in any other research study requiring a special diet, medications, supplements or other lifestyle change

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose and Insulin levels in 1 year as compared to baseline | baseline
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve insulin resistance in subjects with metabolic syndrome. Insulin resistance will be assessed by measuring simultaneously blood glucose and insulin levels in the fasting state and during an oral glucose tolerance test.
Change in Blood Glucose and Insulin levels in 1 year as compared to baseline | after 1 year
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve insulin resistance in subjects with metabolic syndrome. Insulin resistance will be assessed by measuring simultaneously blood glucose and insulin levels in the fasting state and during an oral glucose tolerance test.

SECONDARY OUTCOMES:
Change in abdominal obesity in 1 year as compared to baseline | baseline
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve abdominal obesity and markers of cardiovascular disease in subjects with metabolic syndrome. Abdominal obesity will be measured by both waist circumference and MRI. CVD markers will be measured both in the circulation as well as by MRI estimate of carotid artery intima/media thickness.
Change in abdominal obesity in 1 year as compared to baseline | after 1 year
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve abdominal obesity and markers of cardiovascular disease in subjects with metabolic syndrome. Abdominal obesity will be measured by both waist circumference and MRI. CVD markers will be measured both in the circulation as well as by MRI estimate of carotid artery intima/media thickness.
Change in markers of cardiovascular disease in 1 year as compared to baseline | baseline
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve abdominal obesity and markers of cardiovascular disease in subjects with metabolic syndrome. Abdominal obesity will be measured by both waist circumference and MRI. CVD markers will be measured both in the circulation as well as by MRI estimate of carotid artery intima/media thickness.
Change in markers of cardiovascular disease in 1 year as compared to baseline | after 1 year
  To test whether prolonged (1 year) dietary AGE restriction, while maintaining caloric intake, can improve abdominal obesity and markers of cardiovascular disease in subjects with metabolic syndrome. Abdominal obesity will be measured by both waist circumference and MRI. CVD markers will be measured both in the circulation as well as by MRI estimate of carotid artery intima/media thickness.

CONTACTS AND LOCATIONS:
Overall Officials: John C He, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Uribarri J, Woodruff S, Goodman S, Cai W, Chen X, Pyzik R, Yong A, Striker GE, Vlassara H. Advanced glycation end products in foods and a practical guide to their reduction in the diet. J Am Diet Assoc. 2010 Jun;110(6):911-16.e12. doi: 10.1016/j.jada.2010.03.018. PMID 20497781
- [Background] Mericq V, Piccardo C, Cai W, Chen X, Zhu L, Striker GE, Vlassara H, Uribarri J. Maternally transmitted and food-derived glycotoxins: a factor preconditioning the young to diabetes? Diabetes Care. 2010 Oct;33(10):2232-7. doi: 10.2337/dc10-1058. Epub 2010 Jul 13. PMID 20628088
- [Background] Uribarri J, Cai W, Ramdas M, Goodman S, Pyzik R, Chen X, Zhu L, Striker GE, Vlassara H. Restriction of advanced glycation end products improves insulin resistance in human type 2 diabetes: potential role of AGER1 and SIRT1. Diabetes Care. 2011 Jul;34(7):1610-6. doi: 10.2337/dc11-0091. PMID 21709297
- [Background] Vlassara H, Striker GE. Advanced glycation endproducts in diabetes and diabetic complications. Endocrinol Metab Clin North Am. 2013 Dec;42(4):697-719. doi: 10.1016/j.ecl.2013.07.005. PMID 24286947
- [Background] Striker GE. Beyond phosphate binding: the effect of binder therapy on novel biomarkers may have clinical implications for the management of chronic kidney disease patients. Kidney Int Suppl. 2009 Dec;(114):S1-2. doi: 10.1038/ki.2009.400. No abstract available. PMID 19946321
- [Background] 6. Vlassara, H. and Striker, G.E. (2010) Intake of advanced glycation endproducts; Role in the development of diabetic complications. In: Principles of Diabetes Mellitus, 2nd Edition, L. Poretsky, Ed., Springer Publications.
- [Background] 7. Vlassara, H, Striker, G.E. The Role of AGEs in the Etiology of Insulin Resistance and Diabetes; US-Endocrinology (2011).
- [Derived] Vlassara H, Cai W, Tripp E, Pyzik R, Yee K, Goldberg L, Tansman L, Chen X, Mani V, Fayad ZA, Nadkarni GN, Striker GE, He JC, Uribarri J. Oral AGE restriction ameliorates insulin resistance in obese individuals with the metabolic syndrome: a randomised controlled trial. Diabetologia. 2016 Oct;59(10):2181-92. doi: 10.1007/s00125-016-4053-x. Epub 2016 Jul 29. PMID 27468708